CLINICAL TRIAL: NCT06735456
Title: The Effect of Mandala on Anxiety, Physiological Parameters and Patient Satisfaction in Women With Breast Cancer Receiving Chemotherapy
Brief Title: The Effect of Mandala on Anxiety, Physiological Parameters and Patient Satisfaction in Women With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Filiz Ünal Toprak, Assoc. Prof. Dr., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SBU-FUT-03
Record Dates: First submitted 2024-12-06; First posted 2024-12-16 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Nursing; Mandala
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Two groups with a mandala group and control group
Who Masked: Participant, Outcomes Assessor
Masking Description: Since the application will be performed by the researcher, patients will be blinded in this study. The statistician will be blinded in the evaluation of the data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mandala Group (Experimental): The patient will undergo mandala painting during 1 session of chemotherapy.
  Interventions: Other: Mandala
- Control Group (No Intervention): No application will be made to this group by the researcher.

INTERVENTIONS:
Other: Mandala — The patient will undergo mandala painting during 1 session of chemotherapy.
  Arms: Mandala Group

SUMMARY:
This study will be conducted to examine the effect of mandala painting on anxiety, physiological parameters and patient satisfaction in women with breast cancer receiving chemotherapy.

DETAILED DESCRIPTION:
Breast cancer is among the most common cancers that cause death in women in the world and in our country (1). One of the most commonly used treatment options for breast cancer is chemotherapy. However, many side effects occur depending on the chemotherapy regimen used. The most common side effects in patients receiving chemotherapy are; nausea, vomiting, anemia, fatigue, insomnia, mucositis, and peripheral neuropathy (2, 3). It is stated that the probability of anxiety in people with cancer is 50% or more, while the rate of chronic anxiety is 30%. It is expected that the quality of life will be positively affected by detecting and reducing the level of anxiety and adapting patients to their own treatment (4). Mandala, a type of art therapy method; Although it has various shapes, the round one is generally preferred and is a meditation tool used to convey feelings and thoughts. Studies have shown that art therapy helps individuals feel more peaceful by helping to alleviate strong negative emotions that cause severe discomfort (7). In a study conducted in Hong Kong, the sample group included women with both breast cancer and gynecological cancer. Art therapy was applied to the participants, and as a result of the research, it was observed that the women's psychological distress decreased and their mental well-being increased (8). It is known that the problems experienced by cancer patients can be reduced by changing cognitive focus, similar to art therapy. In a study, cancer patients receiving chemotherapy watched TV series and movies (51.3%), dreamed (26.6%), listened to music (26.6%), visited friends and relatives (19.6%), looked at flowers (14%), walked or walked. It is observed that their depression and anxiety decrease when they engage in activities such as exercising (14%) (9).In the literature, there are mandala studies applied to different patient groups, but no national or international study has been found regarding the effects of mandala painting during chemotherapy in breast cancer patients. Therefore, this study will be conducted to examine the effect of mandala painting on anxiety, physiological parameters and patient satisfaction in women with breast cancer receiving chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with breast cancer,
* Being receiving adjuvant or neoadjuvant chemotherapy,
* Being over 18 years of age,
* Ability to communicate in Turkish,
* Not having a physical disability related to the upper extremities,
* Agreeing to participate in the study.

Exclusion Criteria:

* Advanced stage cancer patients,
* Having visual, hearing and speech disabilities,
* Individuals with mental and neuropsychiatric diseases will not be included in the sample.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Since it is a study conducted on breast cancer women, it concerns the female gender.
Enrollment: 54 (Actual)
Dates: Start 2024-02-24 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Physiological parameter 1 | 2 hours (pre-test and post-test)
  Temperature
Physiological parameter 2 | 2 hours (pre-test and post-test)
  Pulse
Physiological parameter 3 | 2 hours (pre-test and post-test)
  Blood pressure
Physiological parameter 4 | 2 hours (pre-test and post-test)
  spO2
Physiological parameter 5 | 2 hours (pre-test and post-test)
  Respiratory rate

SECONDARY OUTCOMES:
Beck Anxiety Scale | 2 hours (pre-test and post-test)
  The scale is a Likert-type self-evaluation scale consisting of 21 items and scored between 0-3. A high total score indicates the level of anxiety experienced by the person. The score range varies between 0 and 63. Evaluation of the scale is as follows: 0-7 points with no anxiety symptoms, 8-15 with mild anxiety symptoms, 16-25 with moderate anxiety symptoms, and 26-63 with severe anxiety symptoms. Higher scores from the scale mean worse results.

CONTACTS AND LOCATIONS:
Overall Officials: Filiz Ünal Toprak, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Sağlık Bilimleri Üniversitesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No